CLINICAL TRIAL: NCT03176407
Title: Detection of Upper Gastrointestinal (GI) Bleeding With a Novel Bleeding Sensor Capsule: A Pilot Study [DING]
Brief Title: Detection of Upper Gastrointestinal (GI) Bleeding With a Novel Bleeding Sensor Capsule [DING]
Acronym: DING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ovesco Endoscopy AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CT20-HPA-1401
Record Dates: First submitted 2017-04-21; First posted 2017-06-05 (Actual); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: Upper GI Bleeding
Keywords: sensor capsule
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Intervention Model Description: There is only one patient group. The one that swallow the sensor capsule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HemoPill acute (Experimental): Capsule is swallowed by the patient and an external study receiver records the capsule sensor data for 4 consecutive hours.
  Capsule excretion is monitored for up to 4 days. If excretion is not recorded during that time, a follow-up examination of the patient is conducted after 10 days.
  Interventions: Diagnostic Test: HemoPill acute

INTERVENTIONS:
Diagnostic Test: HemoPill acute — Capsule is swallowed by the patient and an external study receiver records the capsule sensor data for 4 consecutive hours. Patients undergo endoscopy within 12 hours after capsule ingestion. Afterwards, the endoscopic findings (endoscopy pictures and patient's endoscopy report) are compared to the sensor capsule data results. Capsule excretion is monitored for up to 4 days. If excretion is not recorded during that time, a follow-up examination of the patient is conducted after 10 days.

SUMMARY:
The clinical trial entitled "Detection of upper gastrointestinal (GI) bleeding with a novel bleeding sensor capsule - a pilot study" was carried out in a monocentric clinical trial with 30 patients. This trial aimed to determine if the capsule's sensor signals allow to deduct the patient's bleeding status in a clinical setting.

The target of the explorative study was to show the feasibility and safety of the HemoPill acute and its implementation procedure as well as, the definition of measurable parameters and thresholds for blood detection. Within this clinical trial, initial clinical data on the performance of the HemoPill acute capsule were collected.

DETAILED DESCRIPTION:
The clinical trial entitled "Detection of upper gastrointestinal (GI) bleeding with a novel bleeding sensor capsule - a pilot study" was carried out in a monocentric clinical trial with 30 patients as part of the final development phase of the HemoPill acute, a bleeding sensor capsule. The swallowable capsule operates with the combination of an optical sensor for blood detection positioned within a recess in the capsule surface and a radio interface for wireless transmission of sensor data to an external receiver device. The HemoPill acute capsule is used for diagnosis of patients with suspected acute upper gastrointestinal bleeding.

For the study, the HemoPill acute capsule was swallowed by the patient and a special extracorporeal receiver was positioned next to the patient's body. The receiver recorded sensor signals from the ingested capsule for the next 4 hours. Patients who had swallowed a capsule underwent endoscopy within the next 12 hours. Later, both the endoscopic pictures and the endoscopy report were compared to the sensor capsule data recorded in the extracorporeal receiver. Furthermore, the excretion of each HemoPill acute capsule was monitored in accordance with the study protocol (regular check to see if sensor signal was still detectable from inside the patient's body) for a follow-up period of 10 days.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion based on anamnestic statements and clinical symptom
* vomiting of hematin (coffee-ground-like material)
* hematemesis
* melena (anamnestic or digital rectal evidence)
* attentive and conscious patient
* written informed consent, age ≥ 18 years and ≤ 80 years

Exclusion Criteria:

* circulatory instability (with a clear need for urgent endoscopy)
* cases which required urgently surgical therapy, e.g. patients previously treated endoscopically because of GI bleeding and with an urgent suspicion of recurrent bleeding, which could not be treated endoscopically because of previous findings as well as patients experiencing re-bleeding after surgery
* known and assumed stenosis of the GI tract, e.g. patients with fistulas, malformations and anatomical variability, insufficiencies, adhesions and previous traumas
* pacemakers or other implantable electrical devices
* difficulties in swallowing pills the size of the capsule known dysphagia (e.g. achalasia, known diverticula of the esophagus etc.) which were inoperable: patients with ASA IV or higher
* known and distinct retardation of the gastro-intestinal tract, induced by previous surgeries, stenosis or paralytic ileus with a diagnosed enteritis
* moribund patient
* pregnancy and breastfeeding
* psychological illnesses, which might impair patient cooperation (comprehension problems, informed consent impossible)
* stomach bezoar
* NSAR-induced enteropathy
* known allergies against Parylene (surface coating of the capsule)
* peptic esophagitis III an IV
* florid M.Crohn or known inflammation-induced strictures
* distinct diverticulosis or diverticulitis
* suspected gastrointestinal tumor disease
* necessity of MRI investigation
* heavy genetic bleeding tendency (e.g. factor VIII deficiency)
* esophagus varices
* class III obesity (BMI ≥ 40)
* missing informed consent
* age < 18 years and > 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04-11 (Actual); Primary Completion 2016-02-24 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gottwald, Prof. Dr., Study Director — Ovesco Endoscopy AG
Locations (1):
- Department of Gastroenterology and Oncology, Klinikum Ludwigsburg, Ludwigsburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmidt A, Zimmermann M, Bauder M, Kuellmer A, Caca K. Novel telemetric sensor capsule for EGD urgency triage: a feasibility study. Endosc Int Open. 2019 Jun;7(6):E774-E781. doi: 10.1055/a-0880-5312. Epub 2019 May 17. PMID 31157295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting to the emergency department with acute UGIB were screened for eligibility. Inclusion criteria were symptoms suggestive of UGIB defined as hematemesis, coffee ground emesis or melena (at least one of three).
Groups:
- HemoPill Acute: There was only one study arm as all patients swallowed the sensor capsule.
Period: Overall Study
Arm/Group | HemoPill Acute
Started | 30
Completed | 27
Not Completed | 3
Not completed — Protocol Violation | 1
Not completed — human failure | 1
Not completed — EGD showed esophageal varices=excl. crit | 1

BASELINE CHARACTERISTICS:
Arm/Group | HemoPill Acute
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants] — Population: Due to the fact that n = 3 dropouts occured.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 8
    >=65 years | 19
Age, Continuous [Mean (Full Range); unit: years] — Population: Due to protocol violations there were n=3 lost to folllow-up patients that were not included in the analysis.
  years | 66 [28 to 80]
Sex: Female, Male [Count of Participants; unit: Participants] — Patients presenting to the emergency department with acute UGIB were screened for eligibility. Inclusion criteria were symptoms suggestive of UGIB defined as hematemesis, coffee ground emesis or melena (at least one of three). Population: Due to protocol violations there were n=3 lost to folllow-up patients that were not included in the analysis.
  Participants
    Female | 10
    Male | 17
Region of Enrollment [Number; unit: participants]
  Germany | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With (Serious) Adverse Event Related to the Medical Device
Description: In this outcome measure the safety of the sensor capsule is evaluated in relation to the patient application.
  1. Every malfunction, failure or characteristic change or performance of the medical device as well as each inappropriate labeling or instruction for use, which can directly or indirectly lead to death or a serious advers event that deteriorates the physical health state of a patient, user or another person.
  2. Every technical or medical reason, which are a result of the causes mentioned in No.1 due to the characteristics or performance of the medical device.
Time Frame: until capsule excretion happened, an average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | HemoPill Acute
Number analyzed (Participants) | 30
Participants | 0

2. Primary Outcome: Number of Participants With Device Deficiencies
Description: All device deficiencies that appear in the study. In this outcome measure the safety and feasibility of the capsule is evaluated.
Time Frame: until data of the receiver is saved, an average of 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HemoPill Acute
Number analyzed (Participants) | 30
Participants | 0

3. Primary Outcome: Number of Participants With Human Failures in Capsule Application
Description: Human failures that appear during the capsule application or data readout.
Time Frame: until capsule excretion happened, an average of 10 days
Population: One human failure occured.
Measure: Count of Participants; unit: Participants
Groups:
- HemoPill Acute: When capsule is swallowed by the patient an external study receiver records the capsule sensor data for 4 consecutive hours.
  After capsule application capsule excretion is monitored for up to 4 days. If excretion is not recorded during that time, a follow-up examination of the patient is conducted after 10 days.
  Capsule readout is performed by the sponsor.
Arm/Group | HemoPill Acute
Number analyzed (Participants) | 30
Participants | 1

4. Primary Outcome: Number of Participants With Sensor Capsule Ingestion Problems
Description: In this outcome measure the feasibility of the capsule is evaluated and if patients have issues on swallowing the sensor capsule in respect to it's size, form or other reasons.
Time Frame: at time of capsule ingestion, 1 day
Measure: Count of Participants; unit: Participants
Groups:
- HemoPill Acute: Capsule is swallowed by the patients themselves. Patient takes the capsule in their hands and put it in their mouth and swallow it by themselves.
Arm/Group | HemoPill Acute
Number analyzed (Participants) | 30
Participants | 0

5. Primary Outcome: Number of Patients Which do Not Accept the Medical Device, Measured in Numbers
Description: Patients that have acceptance problems with the sensor capsule in respect to its size, form or other reasons.
Time Frame: at time of study inclusion, 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | HemoPill Acute
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Arm/Group | HemoPill Acute
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No